CLINICAL TRIAL: NCT03897842
Title: TARGET: A Study to Evaluate the Treatment of Patients With Acute Decompensated Heart Failure (ADHF) Using an Automated Fluid Management System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: CardioRenal Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TARGET0001
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Interventional Arm (Experimental): The initial phase of the study will utilize the Reprieve Cardiovascular System to support a treatment algorithm that maximizes diuretic administration while carefully monitoring patient physiologic and hemodynamic status to ensure safe decongestion.
  Interventions: Device: Reprieve Cardiovascular System

INTERVENTIONS:
Device: Reprieve Cardiovascular System — The Reprieve Cardiovascular System (RCS) shall be utilized to maximize fluid removal over a maximum duration of 72 hours.

SUMMARY:
This is a prospective, single arm, early feasibility study designed to evaluate the safety and device performance of The RenalGuard System in the management of patients admitted with signs and symptoms of congestive heart failure who require diuresis for the treatment of volume overload.

DETAILED DESCRIPTION:
This is a prospective, single arm, early feasibility study designed to evaluate the safety and device performance of The RenalGuard System in the management of patients admitted with signs and symptoms of congestive heart failure who require diuresis for the treatment of volume overload. Subjects will be referred by their physician if he/she feels that the subject could benefit from observed diuresis in a hospital setting.

The device being utilized is called The RenalGuard® System (The System). By default, The System infuses a volume of hydration fluid equal to the volume of urine output. This is known as matched hydration. In addition, the clinician has the ability to adjust the matched setting such that RenalGuard can infuse hydration fluid to achieve a positive fluid balance (e.g. +100 ml/hr.) or a negative fluid balance (e.g. -100 ml/hr.). The purpose of this balanced fluid replacement is to prevent hypovolemia that may lead to hypotension and vital organ dysfunction, or fluid overload that may lead to shortness of breath in subjects in whom high urine output is desired.

All patients will be treated with The RenalGuard System for a minimum of 24-hours, and possibly longer, at the investigators discretion. They will be followed for 30 days post discharge. The protocol will enroll up to 40 subjects to develop the clinical algorithm required to optimally and safely perform removal of volume. The study will be conducted in up to 5 sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Patient ≥18 years old (with body weight ≤160 kg) who is able to provide informed consent
2. Subject is diagnosed and hospitalized with acute decompensated heart failure. ADHF is defined as including all of the following measured at any time between presentation and the end of screening:

   * persistent dyspnea at rest or with minimal exertion at screening and at the time of enrollment, despite standard background therapy for acute heart failure including intravenous furosemide,
   * Rales by chest auscultation
   * Edema ≥ +1 on a 0-3+ scale, indicating indentation of skin with mild digital pressure that requires 10 or more seconds to resolve in any dependent area including extremities or sacral region.
   * pulmonary congestion on chest radiograph
   * systolic BP ≥100 mmHg at the start and at the end of screening
3. Subject with pre-existing chronic renal failure (impaired renal function) defined as an eGFR between presentation and enrollment of ≥ 25 and <90 mL/min/1.73m2, calculated using the MDRD equation.
4. Subject has agreed to all follow-up testing.

Exclusion Criteria:

1. Known inability to have a Foley catheter placed.
2. Total urine output < 200 ml or average urine rate < 50 ml/hour in the Diuretic Challenge.
3. Patient is managed on, or there is a plan to manage on, renal replacement therapy (RRT) such as ultrafiltration, hemofiltration or dialysis.
4. Dyspnea due to non-cardiac causes, such as acute or chronic respiratory disorders or infections (i.e., severe chronic obstructive pulmonary disease, bronchitis, pneumonia), which may interfere with the ability to interpret the primary cause of dyspnea.
5. Patients with blood pressure > 180 mmHg at the time of enrollment or persistent heart rate > 130 bpm.
6. Temperature >38.5°C (oral or equivalent) or sepsis or active infection requiring IV antimicrobial treatment.
7. Clinical evidence of acute coronary syndrome currently or within 30 days prior to enrollment. (Note: the diagnosis of acute coronary syndrome is a clinical diagnosis and that the sole presence of elevated troponin concentrations is not sufficient for a diagnosis of acute coronary syndrome, given that troponin concentrations may be significantly increased in the setting of AHF).
8. AHF due to significant arrhythmias, which include any of the following: sustained ventricular tachycardia or atrial fibrillation/flutter with sustained ventricular response of >130 beats per minute; or bradycardia with sustained ventricular rate <45 beats per minute without the use of a pacemaker
9. Patients with hemoglobin <8 g/dl, or a history of blood transfusion within the 14 days prior to screening, or active life-threatening GI bleeding.
10. Known hepatic impairment (as evidenced by total bilirubin > 3 mg/dL, or increased ammonia levels, if performed) or history of cirrhosis with evidence of portal hypertension such as varices.
11. Significant, uncorrected, left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy or severe aortic stenosis (i.e., aortic valve area <1.0 cm2 or mean gradient >40 mmHg on prior or current echocardiogram) or severe mitral stenosis.
12. Severe aortic insufficiency or severe mitral regurgitation for which surgical or percutaneous intervention is indicated.
13. Documented, prior to or at the time of enrollment, restrictive amyloid myocardiopathy, OR acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy (does NOT include restrictive mitral filling patterns seen on Doppler echocardiographic assessments of diastolic function).
14. Current (within 2 hours prior to enrollment) or planned (through the completion of study drug infusion) treatment with any IV vasoactive therapies, including vasodilators (including nesiritide), positive inotropic agents and vasopressors, or mechanical suport (endotracheal intubation, mechanical ventilation; intra-aortic balloon pump or any ventricular assist device; hemofiltration, ultrafiltration or dialysis), with the exception of IV furosemide (or equivalent diuretic), or IV nitrates at a dose of ≤ 0.1 mg/kg/hour if the patient has a systolic BP >150 mmHg at the start of screening.
15. Any major solid organ transplant recipient or planned/ anticipated organ transplant within 1 year.
16. Major surgery, including implantable devices (e.g. ICD, CRT), or major neurologic event including cerebrovascular events, within 30 days prior to screening.
17. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past year with a current life expectancy less than 1 year due to the malignancy.
18. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
19. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during study treatment plus 5 days after cessation of study treatment.
20. Use of any investigational drugs within 30 days prior to screening.
21. Inability to follow instructions or comply with follow-up procedures.
22. Any other medical condition(s) that may put the patient at risk or influence study results in the investigator's opinion, or that the investigator deems unsuitable for the study, including drug or alcohol abuse or psychiatric, behavioral or cognitive disorders, sufficient to interfere with the patient's ability to understand and comply with the protocol instructions or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
24 Hour Fluid Removal | 24 hours
  The primary efficacy endpoint will be the difference between target fluid loss and actual fluid loss at conclusion of therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Military Hospital of Wroclaw, Wroclaw, Poland